CLINICAL TRIAL: NCT02947152
Title: A Phase I, Multicenter, Open-label Dose Escalation and Expansion Study of HKT288, Administered Intravenously in Adult Patients With Advanced Solid Tumors, Including Epithelial Ovarian Cancer and Renal Cell Carcinoma
Brief Title: HKT288 in Solid Tumors, Including Epithelial Ovarian Cancer and Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHKT288X2101
Record Dates: First submitted 2016-09-12; First posted 2016-10-27 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2018-09

CONDITIONS: Epithelial Ovarian Cancer; Renal Cell Carcinoma
Keywords: HKT288; CDH6; ADC; maytansine; epithelial ovarian cancer; renal cell carcinoma; RCC
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose escalation part (Experimental): Includes patients with serous epithelial ovarian cancer (inclusive of fallopian tubal and peritoneal cancer) and clear cell or papillary renal cell carcinoma
  Interventions: Drug: HKT288
- Dose expansion part (RCC arm) (Experimental): Includes patients with clear cell or papillary renal cell carcinoma
  Interventions: Drug: HKT288
- Dose expansion part (ovarian cancer arm) (Experimental): Includes patients with serous epithelial ovarian cancer (inclusive of fallopian tubal and peritoneal cancer)
  Interventions: Drug: HKT288

INTERVENTIONS:
Drug: HKT288 — Cadherin-6-targeting antibody-drug conjugate for intravenous administration

SUMMARY:
A first-in-human study using HKT288 in solid tumors, including epithelial ovarian cancer and renal cell carcinoma

ELIGIBILITY:
Main Inclusion Criteria:

* Advanced (metastatic or locally advanced) serous epithelial ovarian, serous fallopian tubal or serous primary peritoneal cancer or advanced clear cell or papillary renal cell carcinoma who have received or are intolerant to all therapy known to confer clinical benefit for their disease, as determined by the investigator.
* Tumor sample is available for retrospective CDH6 expression testing
* Eastern Cooperative Oncology Group (ECOG) Performance status ≤2

Main Exclusion Criteria:

* Patient has central nervous system metastatic involvement. Patients with previously treated CNS metastases are also excluded.
* Patient with any active or chronic corneal disorders
* Patients with monocular vision or have media opacities or any other condition that precludes monitoring of the retina or fundus.
* Patients with a history of serious allergic reactions
* Patients with QTcF >470 msec at screening ECG or congenital long QT syndrome
* Any prior history of treatment with maytansine (DM1 or DM4)-based ADC
* Patient have received anti-cancer therapies within the following time frames prior to the first dose of study treatment:

  * Conventional cytotoxic chemotherapy: ≤4 weeks (≤ 6 weeks for nitrosoureas and mitomycin-C)
  * Biologic therapy (e.g., antibodies): ≤4 weeks
  * Non-cytotoxic small molecule therapeutics: ≤5 half-lives or ≤2 weeks (whichever is longer)
  * Other investigational agents: ≤4 weeks
  * Radiation therapy (except for localized radiotherapy for analgesic purpose or for lytic lesions at risk of fracture): ≤4 weeks
  * Radiation therapy (localized radiotherapy for analgesic purpose or for lytic lesions at risk of fracture) ≤2 weeks
  * Major surgery: ≤2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) in the DLT evaluation period | evaluation period is 21 days
Safety assessed by overall incidence of adverse events (AEs) and serious adverse events (SAEs) | Until 105 days after last dose of study treatment (=average of approximately 6 months after first dose)
Tolerability as assessed by numbers of dose changes or interruptions | Until last dose of study treatment (=average of approximately 6 months after first dose)
Safety assessed by severity of adverse events (AEs) and serious adverse events (SAEs) | Until 105 days after last dose of study treatment (=average of approximately 6 months after first dose)

SECONDARY OUTCOMES:
Concentration vs. time profiles of total antibody (tAb) | On treatment up to Cycle 6 Day 1 and at the time of study treatment discontinuation (=average of approximately 6 months after first dose). 1 cycle is 21 days, increases to 28 days if there is a dose delay of 7 days for the start of next dose
Objective response rate | every 2 cycles up to Cycle 17 and every 3 cycles thereafter until study treatment discontinuation (=average of approximately 6 months after first dose). Then every 9 weeks until end of disease progression follow-up (up to 12 months)
Duration of response | every 2 cycles up to Cycle 17 and every 3 cycles thereafter until study treatment discontinuation (=average of approximately 6 months after first dose). Then every 9 weeks until end of disease progression follow-up (up to 12 months)
Progression-free survival | every 2 cycles up to Cycle 17 and every 3 cycles thereafter until study treatment discontinuation (=average of approximately 6 months after first dose). Then every 9 weeks until end of disease progression follow-up (up to 12 months)
Disease Control Rate | At 6 months on treatment
Best overall response | every 2 cycles up to Cycle 17 and every 3 cycles thereafter until study treatment discontinuation (=average of approximately 6 months after first dose). Then every 9 weeks until end of disease progression follow-up (up to 12 months)
Presence of anti-HKT288 antibodies. | On treatment up to Cycle 6 Day 1 and at the time of study treatment discontinuation (=average of approximately 6 months after first dose)
CDH6 expression level | 3 months
Pharmacokinetics (PK) parameter (AUC) for HKT288 | On treatment up to Cycle 6 Day 1 and at the time of study treatment discontinuation (=average of approximately 6 months after first dose)
PK parameter (Cmax) for HKT288 | On treatment up to Cycle 6 Day 1 and at the time of study treatment discontinuation (=average of approximately 6 months after first dose)
PK parameter (Tmax) for HKT288 | On treatment up to Cycle 6 Day 1 and at the time of study treatment discontinuation (=average of approximately 6 months after first dose)
PK parameters (half-life) for HKT288 | On treatment up to Cycle 6 Day 1 and at the time of study treatment discontinuation (=average of approximately 6 months after first dose)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Novartis Investigative Site, Houston, Texas, United States
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Nagoya, Aichi-ken, Japan
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Locarno, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CHKT288X2101 can be found on the Novartis Clinical Trials Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17224